CLINICAL TRIAL: NCT05897476
Title: Prospective Feasibility Study of Point-of-care Ultrasound in Suspected Aortic Dissection
Acronym: FESDAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/781
Record Dates: First submitted 2023-05-26; First posted 2023-06-09 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2023-05

CONDITIONS: Aortic Dissection; Emergency Ultrasound
MeSH Terms: conditions — Aortic Dissection | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Prospective single-center interventional diagnostic
  H1: inclusion interview then :
  Medical interrogation (retrospective collection if already done / but additional requests if missing data).
  Clinical examination (complementary if missing data).
  Ultrasound with 3 ultrasound sections to be performed: parasternal long axis, supra-sternal and abdominal, looking for the following signs:
  Direct signs: presence of an intimal flap, intramural aortic hematoma > 5mm, penetrating aortic ulcer.
  Indirect signs: pericardial effusion, aortic dilatation ≥ 4 cm, tamponade (1). H4: retrospective collection of the results of complementary examinations if any, biological and radiological, and collection of the final diagnosis retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultrasound arm (Experimental): every patient will be examine with ultrasound
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound — brief external ultrasound will be proceed on each patient included searching signs of aortic dissection

SUMMARY:
Aortic dissection is an uncommon and serious pathology. Its diagnosis is difficult because of the varied and silent clinical presentations. The development of ultrasound in emergency medicine is an asset in certain pathologies. The aim of this study is therefore to study the feasibility of a protocol integrating clinical ultrasound in the suspicion of acute aortic dissection in the hospital setting. This study is a single-center prospective interventional study. In which the investigators perform ultrasound in patients with suspected acute aortic dissection in the emergency department. If the protocol is feasible and if it allows a saving of time in the diagnosis or an increase in diagnoses, the investigators will be able to evoke a profitability to the systematic realization of this examination.

DETAILED DESCRIPTION:
H0: patient selection and inclusion:

* Presentation of the study
* Delivery of the information note / no objection to the patient if he/she is in a state to consent
* Emergency procedure:

In accordance with article L-1122-1-3 of the public health code, patients may be included in the study at the initiative of the physician without seeking prior consent. This procedure will be associated with a prior call to the relatives to obtain an oral consent in principle (traced in the patient's medical file), while waiting for the delivery of the information note / no objection to the relatives and then to the patient as soon as his condition allows it.

H1: inclusion interview then :

Medical interrogation (retrospective collection if already done / but additional requests if missing data).

Clinical examination (complementary if missing data).

Ultrasound with 3 ultrasound sections to be performed: parasternal long axis, supra-sternal and abdominal, looking for the following signs:

Direct signs: presence of an intimal flap, intramural aortic hematoma > 5mm, penetrating aortic ulcer.

Indirect signs: pericardial effusion, aortic dilatation ≥ 4 cm, tamponade (1).

H4: retrospective collection of the results of complementary examinations if any, biological and radiological, and collection of the final diagnosis retained.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-95 years included
* Non-opposition of the subject to participate in the study
* All patients admitted to the emergency department of the Besançon University Hospital With chest, abdominal, back, lumbar pain, or acute headache
* AORTA score ≥ 1
* Clinical suspicion of AD by the emergency physician

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate with the study and/or poor cooperation anticipated by the investigator
* Subject without health insurance
* Pregnant woman
* ECG showing acute coronary syndrome and/or ventricular rhythm disturbances
* Traumatic context, or traumatic cause of pain
* Chronic / subacute dissection (patient with incidental discovery of aortic dissection (city assessment) and then referred to the emergency room).
* Patient refusal to participate in the study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2023-12-24 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Successful completion of FESDAU protocol. | 15 minutes
  The statistical analysis on the primary endpoint will be a percentage of success in completing the FESDAU protocol among all eligible individuals.

SECONDARY OUTCOMES:
time to diagnosis | 24 hours
  time to diagnosis with FESDAU protocol
Time to perform the ultrasound | 60 minutes
  during of processing ultrasound
Ultrasound slices with a suggestive sign | 60 minutes
  wich slices are the most interesting

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Besancon, Besançon, France